CLINICAL TRIAL: NCT02021955
Title: Integrating Care After Exacerbation of COPD (InCasE)
Brief Title: Integrating Care After Exacerbation of COPD
Acronym: InCasE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 12-130
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Results first posted 2021-06-04 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: randomized controlled trial; quality of life; patient readmission; mortality; patient satisfaction; intervention studies; multicenter study
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- usual care (No Intervention): Primary care providers treat their patients discharged from hospital for a COPD exacerbation as usual.
- guideline treatment recommendations (Experimental): Primary care clinicians receive treatment recommendations for their patients discharged from hospital for a COPD exacerbation.
  Interventions: Behavioral: guideline treatment recommendations

INTERVENTIONS:
Behavioral: guideline treatment recommendations — Primary care clinicians receive guideline concordant treatment recommendations for their patients discharged from hospital for a COPD exacerbation.
  Arms: guideline treatment recommendations

SUMMARY:
This clinical trial is designed to determine whether an intervention that provides information to primary care providers about gaps in care for their patients recently discharged from hospital for COPD can reduce hospital re-admissions and mortality and improve their patients' quality-of-life.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) exacerbations are common among Veterans admitted to hospital, lead to worsening health-related quality of life, and are important drivers of health care expenditures. As many as half of patients discharged for COPD are readmitted within 6 months. An intervention to improve COPD care is needed, not only to treat patients for COPD and their accompanying comorbidities, but also to redesign the care delivery system. The goal of this clinical trial is to test an intervention to improve patient care during the transition from hospital to outpatient setting for patients discharged for COPD. The investigators are targeting the intervention to Patient Aligned Care Team (PACT) providers who are randomized to receive the intervention or not receive the intervention. For the intervention, study clinicians, consisting of experienced primary care providers and pulmonary specialists, reviewed the medical record for each patient discharged from hospital for COPD. The team looked for gaps in care for COPD and key co-morbidities such as obesity, hypertension, diabetes, and cardiovascular disease. They focused on immediate care processes associated with the hospital admission and comorbid disease treatment. For providers in the intervention group, the team placed any patient care recommendations into the medical record using a non-visit consult note and pre-filled order sets. The patient's provider then accepted, modified, or declined any or all of the recommendations based on personal knowledge of the patient's history. The investigators hypothesize that the intervention will: 1) improve patient quality of life; and 2) decrease hospital readmission and mortality after hospital admission for COPD exacerbation.

ELIGIBILITY:
Inclusion Criteria:

Providers:

* Primary care provider (MD, NP, PA) from VA Puget Sound or Boise VA.
* Willingness to participate in the informed consent process and complete interviews and questionnaires.

Patients:

* Having a provider that is participating in this clinical trial.
* Discharged alive with either a primary discharge diagnosis of COPD or acute respiratory failure with a secondary diagnosis of COPD.
* Willing and able to participate in the informed consent process and complete interviews and questionnaires.

Exclusion Criteria:

Providers: none

Patients:

* Having previously participated in the study.
* Significant cognitive dysfunction, language barrier, or severe psychiatric disorder that would preclude completing the questionnaires.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 717 (Actual)
Dates: Start 2015-02-11 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H. Au, MD MS, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (2):
- United States (2):
  - Boise VA Medical Center, Boise, ID, Boise, Idaho
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Au DH, Collins MP, Berger DB, Carvalho PG, Nelson KM, Reinke LF, Goodman RB, Adamson R, Woo DM, Rise PJ, Coggeshall SS, Plumley RB, Epler EM, Moss BR, McDowell JA, Weppner WG. Health System Approach to Improve Chronic Obstructive Pulmonary Disease Care after Hospital Discharge: Stepped-Wedge Clinical Trial. Am J Respir Crit Care Med. 2022 Jun 1;205(11):1281-1289. doi: 10.1164/rccm.202107-1707OC. PMID 35333140

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We grouped primary care teams into 30 clusters and randomly assigned each cluster to one of 30 30-day time periods at which time the team would moved from control to intervention. Teams gained and lost providers each month as indicated by addition and attrition below. We also have indicated the number of eligible patient discharges that occurred for each group.
Pre-assignment Details: Prior to randomization, 224 providers were invited with 7 refusing, leaving 217 providers included in randomization; 7 additional providers left primary care prior to Step 0, leaving 210 providers who initially participated in the control group in Step 0.
Units Other Than Participants: Clusters of primary care providers
Period: Step 0
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 210; 30 Clusters of primary care providers (Provider attrition=2; Provider addition=3; Patient discharges=14) | 0; 0 Clusters of primary care providers (Provider attrition=0; Provider addition=0; Patient discharges=0)
Completed | 210; 30 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 1
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 193; 29 Clusters of primary care providers (Provider attrition=20; Provider addition=2; Patient discharges=14) | 18; 1 Clusters of primary care providers (Provider attrition=7; Provider addition=0; Patient discharges: 0)
Completed | 193; 29 Clusters of primary care providers | 18; 1 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 2
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 165; 28 Clusters of primary care providers (Provider attrition=5; Provider addition=21; Patient discharges=12) | 21; 2 Clusters of primary care providers (Provider attrition=2; Provider addition=5; Patient discharges=2)
Completed | 165; 28 Clusters of primary care providers | 21; 2 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 3
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 175; 27 Clusters of primary care providers (Provider attrition=2; Provider addition=4; Patient discharges=5) | 30; 3 Clusters of primary care providers (Provider attrition=0; Provider addition=3; Patient discharges=3)
Completed | 175; 27 Clusters of primary care providers | 30; 3 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 4
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 173; 26 Clusters of primary care providers (Provider attrition=0; Provider addition=3; Patient discharges: 13) | 37; 4 Clusters of primary care providers (Provider attrition=0; Provider addition=1; Patient discharges=0)
Completed | 173; 26 Clusters of primary care providers | 37; 4 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 5
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 174; 25 Clusters of primary care providers (Provider attrition=3; Provider addition=0; Patient discharges=11) | 40; 5 Clusters of primary care providers (Provider attrition=0; Provider addition=0; Patient discharges=2)
Completed | 174; 25 Clusters of primary care providers | 40; 5 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 6
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 158; 24 Clusters of primary care providers (Provider attrition=0; Provider addition=2; Patient discharges=6) | 53; 6 Clusters of primary care providers (Provider attrition=0; Provider addition=1; Patient discharges=1)
Completed | 158; 24 Clusters of primary care providers | 53; 6 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 7
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 157; 23 Clusters of primary care providers (Provider attrition=0; Provider addition=2; Patient discharges=13) | 57; 7 Clusters of primary care providers (Provider attrition=0; Provider addition=1; Patient discharges=2)
Completed | 157; 23 Clusters of primary care providers | 57; 7 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 8
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 144; 22 Clusters of primary care providers (Provider attrition=1; Provider addition=0; Patient discharges=9) | 73; 8 Clusters of primary care providers (Provider attrition=0; Provider addition=0; Patient discharges=11)
Completed | 144; 22 Clusters of primary care providers | 73; 8 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 9
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 139; 21 Clusters of primary care providers (Provider attrition=2; Provider addition=1; Patient discharges=9) | 77; 9 Clusters of primary care providers (Provider attrition=1; Provider addition=0; Patient discharges=8)
Completed | 139; 21 Clusters of primary care providers | 77; 9 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 10
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 135; 20 Clusters of primary care providers (Provider attrition=0; Provider addition=1; Patient discharges: 8) | 79; 10 Clusters of primary care providers (Provider attrition=1; Provider addition=0; Patient discharges=5)
Completed | 135; 20 Clusters of primary care providers | 79; 10 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 11
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 126; 19 Clusters of primary care providers (Provider attrition=1; Provider addition=0; Patient discharges=11) | 88; 11 Clusters of primary care providers (Provider attrition=2; Provider addition=2; Patient discharges=7)
Completed | 126; 19 Clusters of primary care providers | 88; 11 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 12
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 123; 18 Clusters of primary care providers (Provider attrition=1; Provider addition=0; Patient discharges=3) | 90; 12 Clusters of primary care providers (Provider attrition=0; Provider addition=2; Patient discharges=1)
Completed | 123; 18 Clusters of primary care providers | 90; 12 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 13
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 118; 17 Clusters of primary care providers (Provider attrition=10; Provider addition=0; Patient discharges=4) | 96; 13 Clusters of primary care providers (Provider attrition=4; Provider addition=0; Patient discharges=5)
Completed | 118; 17 Clusters of primary care providers | 96; 13 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 14
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 105; 16 Clusters of primary care providers (Provider attrition=1; Provider addition=9; Patient discharges=7) | 95; 14 Clusters of primary care providers (Provider attrition=7; Provider addition=11; Patient discharges=3)
Completed | 105; 16 Clusters of primary care providers | 95; 14 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 15
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 110; 15 Clusters of primary care providers (Provider attrition=0; Provider addition=0; Patient discharges=4) | 102; 15 Clusters of primary care providers (Provider attrition=0; Provider addition=5; Patient discharges=5)
Completed | 110; 15 Clusters of primary care providers | 102; 15 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 16
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 103; 14 Clusters of primary care providers (Provider attrition=0; Provider addition=0; Patient discharges=2) | 114; 16 Clusters of primary care providers (Provider attrition=0; Provider addition=3; Patient discharges=3)
Completed | 103; 14 Clusters of primary care providers | 114; 16 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 17
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 99; 13 Clusters of primary care providers (Provider attrition=0; Provider addition=0; Patient discharges=8) | 121; 17 Clusters of primary care providers (Provider attrition=0; Provider addition=0; Patient discharges=3)
Completed | 99; 13 Clusters of primary care providers | 121; 17 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 18
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 96; 12 Clusters of primary care providers (Provider attrition=0; Provider addition=0; Patient discharges=6) | 124; 18 Clusters of primary care providers (Provider attrition=0; Provider addition=0; Patient discharges=7)
Completed | 96; 12 Clusters of primary care providers | 124; 18 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 19
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 94; 11 Clusters of primary care providers (Provider attrition=0; Provider addition=0; Patient discharges=5) | 126; 19 Clusters of primary care providers (Provider attrition=0; Provider addition=0; Patient discharges=9)
Completed | 94; 11 Clusters of primary care providers | 126; 19 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 20
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 92; 10 Clusters of primary care providers (Provider attrition=0; Provider addition=1; Patient discharges=9) | 128; 20 Clusters of primary care providers (Provider attrition=0; Provider addition=1; Patient discharges=9)
Completed | 92; 10 Clusters of primary care providers | 128; 20 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 21
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 88; 9 Clusters of primary care providers (Provider attrition=0; Provider addition=7; Patient discharges=1) | 134; 21 Clusters of primary care providers (Provider attrition=0; Provider addition=12; Patient discharges=9)
Completed | 88; 9 Clusters of primary care providers | 134; 21 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 22
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 89; 8 Clusters of primary care providers (Provider attrition=0; Provider addition=0; Patient discharges=8) | 152; 22 Clusters of primary care providers (Provider attrition=0; Provider addition=3; Patient discharges=8)
Completed | 89; 8 Clusters of primary care providers | 152; 22 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 23
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 69; 7 Clusters of primary care providers (Provider attrition=0; Provider addition=1; Patient discharges=3) | 175; 23 Clusters of primary care providers (Provider attrition=0; Provider addition=0; Patient discharges=7)
Completed | 69; 7 Clusters of primary care providers | 175; 23 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 24
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 62; 6 Clusters of primary care providers (Provider attrition=0; Provider addition=0; Patient discharges=4) | 183; 24 Clusters of primary care providers (Provider attrition=1; Provider addition=1; Patient discharges=8)
Completed | 62; 6 Clusters of primary care providers | 183; 24 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 25
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 37; 5 Clusters of primary care providers (Provider attrition=0; Provider addition=1; Patient discharges=0) | 208; 25 Clusters of primary care providers (Provider attrition=1; Provider addition=0; Patient discharges=5)
Completed | 37; 5 Clusters of primary care providers | 208; 25 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 26
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 30; 4 Clusters of primary care providers (Provider attrition=0; Provider addition=0; Patient discharges=2) | 215; 26 Clusters of primary care providers (Provider attrition=0; Provider addition=23; Patient discharges=9)
Completed | 30; 4 Clusters of primary care providers | 215; 26 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 27
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 25; 3 Clusters of primary care providers (Provider attrition=1; Provider addition=1; Patient discharges=0) | 243; 27 Clusters of primary care providers (Provider attrition=1; Provider addition=4; Patient discharges=4)
Completed | 25; 3 Clusters of primary care providers | 243; 27 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 28
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 15; 2 Clusters of primary care providers (Provider attrition=0; Provider addition=2; Patient discharges=0) | 256; 28 Clusters of primary care providers (Provider attrition=3; Provider addition=6; Patient discharges=6)
Completed | 15; 2 Clusters of primary care providers | 256; 28 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 29
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 10; 1 Clusters of primary care providers (Provider attrition=0; Provider addition=0; Patient discharges=0) | 266; 29 Clusters of primary care providers (Provider attrition=1; Provider addition=2; Patient discharges=8)
Completed | 10; 1 Clusters of primary care providers | 266; 29 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers
Period: Step 30
Arm/Group | Usual Care | Guideline Treatment Recommendations
Started | 0; 0 Clusters of primary care providers (Provider attrition=0; Provider addition=0; Patient discharges=0) | 277; 30 Clusters of primary care providers (Provider attrition=0; Provider addition=1; Patient discharges=11)
Completed | 0; 0 Clusters of primary care providers | 277; 30 Clusters of primary care providers
Not Completed | 0; 0 Clusters of primary care providers | 0; 0 Clusters of primary care providers

BASELINE CHARACTERISTICS:
Groups:
- Provider Participants: all primary care providers: demographic information not collected
- Control Patient Participants: data for all patients discharged under care of a provider in the control group
- Intervention Patient Participants: data for all patients discharged under care of a provider in the intervention group
- Total: Total of all reporting groups
Arm/Group | Provider Participants | Control Patient Participants | Intervention Patient Participants | Total
Number analyzed (Participants) | 365 | 191 | 161 | 717
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Demographic information not collected from provider participants
  years
    number analyzed (Participants) | 0 | 191 | 161 | 352
    (all) |  | 69.7 (8.6) | 69.7 (8.1) | 69.7 (8.35)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Demographic information not collected for provider participants
  Participants
    number analyzed (Participants) | 0 | 191 | 161 | 352
    Female |  | 182 | 155 | 337
    Male |  | 9 | 6 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Demographic information not collected from provider participants
  Participants
    number analyzed (Participants) | 0 | 191 | 161 | 352
    American Indian or Alaska Native |  | 1 | 3 | 4
    Asian |  | 2 | 3 | 5
    Native Hawaiian or Other Pacific Islander |  | 0 | 5 | 5
    Black or African American |  | 8 | 14 | 22
    White |  | 166 | 120 | 286
    More than one race |  | NA — not collected | NA — not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
    Unknown or Not Reported |  | 14 | 16 | 30
Provider type [Number; unit: provider participants] — Population: Data are for those providers that had at least one patient discharged for COPD within the intervention period
  provider participants
    Nurse Practitioner/Physician Assistant: number analyzed (Participants) | 139 | 0 | 0 | 139
    Nurse Practitioner/Physician Assistant | 38 |  |  | 38
    Attending Physician: number analyzed (Participants) | 139 | 0 | 0 | 139
    Attending Physician | 66 |  |  | 66
    Physician Fellow/Resident Physician: number analyzed (Participants) | 139 | 0 | 0 | 139
    Physician Fellow/Resident Physician | 35 |  |  | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Hospital Re-admission and Mortality
Description: Composite measure of hospital readmission for any cause at 180 days and all-cause mortality.
Time Frame: 180 days post-discharge
Population: For 365 enrolled providers, we analyzed 352 patients discharged from hospital for COPD for readmission or mortality
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Guideline Treatment Recommendations
Number analyzed (Participants) | 191 | 161
Participants | 84 | 61

2. Primary Outcome: COPD-related Patient Quality-of-life (Clinical COPD Questionnaire)
Description: self-report survey of patients' quality-of-life with scores ranging from 0-6 with lower scores representing better health; not all participants completed surveys.
Time Frame: 6 weeks post-discharge
Population: For 365 enrolled providers, we surveyed 352 patients discharged from hospital for COPD. Not all participants completed surveys.
Measure: Mean (Standard Deviation); unit: CCQ total score
Arm/Group | Usual Care | Guideline Treatment Recommendations
Number analyzed (Participants) | 97 | 70
CCQ total score | 3.50 (1.22) | 2.97 (1.20)

3. Secondary Outcome: Patients Participants' General Health Status (Veterans RAND 12 Item Health Survey ) Physical Component Score (VR-12 PCS)
Description: self-report survey of patients' general physical health quality-of-life scored from 0-100 with higher scores indicating better health.
Time Frame: 6 weeks post-discharge
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Guideline Treatment Recommendations
Number analyzed (Participants) | 88 | 62
units on a scale | 29.92 (12.22) | 33.25 (11.94)

ADVERSE EVENTS:
Time Frame: 180 days after index hospital discharge
Description: Systematic adverse event review occurred after a patient's 180-day outcomes period when a coordinator reviewed the electronic health record (EHR) for pertinent events.
  Adverse events were not collected for provider participants. Adverse events are reported only for patient participants.
Arm/Group | Usual Care | Guideline Treatment Recommendations
All-Cause Mortality (participants affected / at risk) | 21/191 | 15/161
Serious Adverse Events (participants affected / at risk) | 84/191 | 68/161
Other Adverse Events (participants affected / at risk) | 20/191 | 38/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=191) | Guideline Treatment Recommendations (N=161)
Overall number (General disorders) | 84 (152) | 68 (115) — Adverse events not collected at body system level; collected only at the general level
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=191) | Guideline Treatment Recommendations (N=161)
Non-serious Adverse events (General disorders) | 20 (34) | 38 (104) — AEs not collected at body system level; collected only at the general level

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT02021955/Prot_SAP_000.pdf